CLINICAL TRIAL: NCT04662489
Title: Radial Ablation for the Control of Persistent Atrial Fibrillation (Ablación Radial Para conTrol de la fibrilación Auricular persISTtente)
Brief Title: Radial Ablation for the Control of Persistent Atrial Fibrillation
Acronym: ARTIST
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Innovacion en Biomedicina (FIBMED) (Other)
Collaborators: Hospital General Universitario Gregorio Marañon (Other); Hospital Universitario 12 de Octubre (Other); Puerta de Hierro University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARTIST
Record Dates: First submitted 2020-11-24; First posted 2020-12-10 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Persistent Atrial Fibrillation
Keywords: Atrial fibrillation; Catheter ablation; Radial ablation; Rotors
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Control and treatment arms. Control group refers to pulmonary vein isolation ablation. Treatment group refers to pulmonary vein isolation plus radial ablation of rotational activity sites.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control arm. Pulmonary vein isolation (Active Comparator): Pulmonary vein isolation with ablation.
  Interventions: Procedure: Pulmonary vein electrical isolation
- Treatment arm. Radial ablation (Experimental): Pulmonary vein isolation plus radial ablation of rotational activity sites.
  Interventions: Procedure: Radial ablation

INTERVENTIONS:
Procedure: Pulmonary vein electrical isolation — Electrical isolation of the pulmonary veins from the left atrium with cryoablation therapy
  Other Names: Pulmonary veins ablation
  Arms: Control arm. Pulmonary vein isolation
Procedure: Radial ablation — Electrical isolation of the pulmonary veins from the left atrium plus radial ablation of rotational activity sites with radiofrequency ablation.
  Arms: Treatment arm. Radial ablation

SUMMARY:
The protocol aims to evaluate the efficacy of the radial ablation technique of the maintenance mechanisms in persistent atrial fibrillation compared to the isolation of the pulmonary veins evaluating the atrial fibrillation burden during one year follow-up.

DETAILED DESCRIPTION:
Atrial fibrillation is the most common arrhythmia in clinical practice, and its treatment still remains suboptimal. Electrical isolation of the pulmonary veins with radiofrequency ablation or cryoablation is the standard therapy when antiarrhythmic drugs or electrical cardioversion is not successful. However, recurrence after catheter ablation worsens in persistent and permanent atrial fibrillation patients. Recently, rotational activity electrogram patterns of self-sustained electrical activity found in the atria have been proposed as the responsible mechanism for the maintenance of atrial fibrillation. The investigators devised a controlled, multicentric, prospective, not blinded, and randomized clinical trial with the aim of comparing pulmonary vein catheter ablation versus radial ablation of sites exhibiting rotational activity in patients with persistent atrial fibrillation. Radial ablation consists of the ablation of the rotational activity sites and an additional ablation line connecting the rotation site with the circumferential ablation line of the pulmonary veins.

Besides, subanalysis ARTIST-Gender and ARTIST-HF will be performed. ARTIST-Gender will compare the same outcomes and analysis of the patient cohort but according to the gender of the patient, and ARTIST-HF will sub-divide the analysis with respect to heart failure present in the enrolled patients' cohort.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤ 75 years.
* Non-valvular symptomatic persistent atrial fibrillation.
* Patient willingness to participate in the study providing signed written informed consent.
* Failure or drug intolerance or refusal to continue with chronic antiarrhythmic treatment.
* Left ventricular ejection fraction LVEF) ≥ 25 % in the last echocardiogram prior to enrollment.

Exclusion Criteria:

* Left atrial diameter > 5.5 cm in the last echocardiogram.
* Contraindication of chronic anticoagulation or heparin.
* Previous atrial fibrillation ablation procedure.
* Acute coronary syndrome, cardiac surgery or acute cerebrovascular accident in two months prior to enrollement.
* Previous diagnosis for hyperthyroidism or hypothyroidism.
* Mental or physical illness that disables the patient to participate in the study.
* Scheduled cardiac percutaneous or surgical intervention.
* Non-controlled hypertension > 160/100.
* Terminal renal insufficiency or dialysis.
* Functional class IV of the New York Heart Association (NYHA).
* Moderate valvular disease or previous mitral prosthesis.
* Previous hypertrophic heart disease.
* Life expectancy less than 12 months.
* Inclusion on the transplant list.
* Participation in another study so as not to interfere with the results.
* Previous atrioventricular block.
* Pericardial effusion.
* Pregnancy or childbearing age without contraceptive treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation burden (1 year) | Patients will be followed up during one year, regardless of reaching or not the primary endpoint.
  Atrial fibrillation burden. Holter monitoring at 4, 8 and 12 months. Time to first atrial fibrillation episode.
  Extended analyses by gender and heart failure presence in subanalyses ARTIST-Gender and ARTIST-HF.
Atrial flutter burden (1 year) | Patients will be followed up during one year, regardless of reaching or not the primary endpoint.
  Atrial flutter burden. Holter monitoring at 4, 8 and 12 months. Time to first atrial flutter episode.
  Extended analyses by gender and heart failure presence in subanalyses ARTIST-Gender and ARTIST-HF.
Atrial tachycardia burden (1 year) | Patients will be followed up during one year, regardless of reaching or not the primary endpoint.
  Atrial tachycardia burden. Holter monitoring at 4, 8 and 12 months. Time to first atrial tachycardia episode.
  Extended analyses by gender and heart failure presence in subanalyses ARTIST-Gender and ARTIST-HF.

SECONDARY OUTCOMES:
Occurrence of severe complication of the ablation procedure | 2 years
  Occurrence of severe complications of the ablation procedure Will be identified through review of patient clinical reports. One week post-procedural complications included.
  Extended analyses by gender and heart failure presence in subanalyses ARTIST-Gender and ARTIST-HF.
Overall clinical procedure, radiofrequency and fluoroscopy durations | 2 years
  Total time registered during the clinical procedure.
  Extended analyses by gender and heart failure presence in subanalyses ARTIST-Gender and ARTIST-HF.
Accute procedural success rate | 2 years
  Accute procedural success as the percentage of episodes that revert to sinus flutter or sinus rhythm during the ablation procedure.
  Extended analyses by gender and heart failure presence in subanalyses ARTIST-Gender and ARTIST-HF.
Occurrence of hospitalization for cardiovascular cause | 1 year
  Unforeseen hospitalization for cardiovascular cause requiring overnight hospital stay during the 12 month follow-up.
  Extended analyses by gender and heart failure presence in subanalyses ARTIST-Gender and ARTIST-HF.
Cerebrovascular accident unforeseen hospitalization | 1 year
  Unforeseen hospitalization due to cerebrovascular accident (CVA) requiring overnight hospital stay during the 12 month follow-up.
  Extended analyses by gender and heart failure presence in subanalyses ARTIST-Gender and ARTIST-HF.
Heart failure unforeseen hospitalization | 1 year
  Unforeseen hospitalization due to new diagnosis for heart failure requiring overnight hospital stay during the 12 month follow-up.
  Extended analyses by gender and heart failure presence in subanalyses ARTIST-Gender and ARTIST-HF.
Functional class worsening unforeseen hospitalization | 1 year
  Unforeseen hospitalization due to functional class worsening due to heart failure requiring overnight hospital stay during the 12 month follow-up.
  Extended analyses by gender and heart failure presence in subanalyses ARTIST-Gender and ARTIST-HF.
Final functional class at the end of the study | 2 years
  Final functional class at the end of the study. New York Heart Association (NYHA) classification.
  Extended analyses by gender and heart failure presence in subanalyses ARTIST-Gender and ARTIST-HF.
Total and cardiac mortality | 2 years
  Total and cardiac mortality
  Extended analyses by gender and heart failure presence in subanalyses ARTIST-Gender and ARTIST-HF.
Quality of life measured with the The Short Form (36) Health Survey | 1 year
  Quality of life is measured with the The Short Form (36) Health Survey at pre-specified study follow-up visits (4, 8, 12 months).
  The short-form (36) health survey consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
  Extended analyses by gender and heart failure presence in subanalyses ARTIST-Gender and ARTIST-HF.

CONTACTS AND LOCATIONS:
Overall Officials: Angel Arenal, MD, PhD, Principal Investigator — Hospital General Universitario Gregorio Marañón
Locations (3):
- Spain (3):
  - Hospital General Universitario Gregorio Marañon, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid

IPD SHARING:
Plan to Share IPD: No